CLINICAL TRIAL: NCT04502602
Title: A Phase 1/1b Clinical Trial of Niraparib and Neratinib in Advanced Solid Tumors With an Expansion Cohort in Platinum-resistant Ovarian Cancer
Brief Title: Niraparib and Neratinib in Advanced Solid Tumors With Expansion Cohort in Advanced Ovarian Cancer
Acronym: iNNOVATE
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Puma Biotechnology, Inc. (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18-14152; NCI-2020-05315 (Other: NCI CTRP)
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Advanced Solid Tumor; Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — neratinib; niraparib

STUDY DESIGN:
Intervention Model Description: Dose escalation will proceed within each cohort. Phase 1b is the expansion cohort at the recommended phase 2 dose found in phase 1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Dose Level -1 (Experimental): Neratinib 160 mg and Niraparib 100 mg by mouth once daily for 28 day cycles.
  Interventions: Drug: Neratinib 160 mg; Drug: Niraparib 100 mg
- Dose Level 1 (Experimental): Neratinib 160 mg and Niraparib 200 mg by mouth once daily for 28 day cycles.
  Interventions: Drug: Neratinib 160 mg; Drug: Niraparib 200 mg
- Dose Level 2 (Experimental): Neratinib 200 mg and Niraparib 200 mg by mouth once daily for 28 day cycles.
  Interventions: Drug: Neratinib 200 mg; Drug: Niraparib 200 mg
- Dose Level 3 (Experimental): Neratinib 240 mg and Niraparib 200 mg by mouth once daily for 28 day cycles.
  Interventions: Drug: Neratinib 240 mg; Drug: Niraparib 200 mg
- Dose Level 4 (Experimental): Neratinib 240 mg and Niraparib 300 mg by mouth once daily for 28 day cycles.
  Interventions: Drug: Neratinib 240 mg; Drug: Niraparib 300 mg
- Phase 1b: Platinum Resistant Expansion Cohort (Experimental): This portion of the study provides for cohort expansion to observe for 4 month or greater progression-free survival in patients with platinum resistant ovarian cancer treated at the recommended phase 2 dose (RP2D) determined in Phase I.
  Interventions: Drug: Niraparib at RP2D; Drug: Neratinib at RP2D

INTERVENTIONS:
Drug: Neratinib 160 mg — Escalating doses to determine recommended phase 2 dose (RP2D)
  Arms: Dose Level -1; Dose Level 1
Drug: Neratinib 200 mg — Determined RP2D dose
  Arms: Dose Level 2
Drug: Neratinib 240 mg — Escalating doses to determine recommended phase 2 dose (RP2D)
  Arms: Dose Level 3; Dose Level 4
Drug: Niraparib 100 mg — Escalating doses to determine recommended phase 2 dose (RP2D)
  Arms: Dose Level -1
Drug: Niraparib 200 mg — Escalating doses to determine recommended phase 2 dose (RP2D)
  Arms: Dose Level 1; Dose Level 2; Dose Level 3
Drug: Niraparib 300 mg — Phase 1: Escalating doses to determine recommended phase 2 dose (RP2D)
  Arms: Dose Level 4
Drug: Niraparib at RP2D — Phase 1b: Determined dose
  Arms: Phase 1b: Platinum Resistant Expansion Cohort
Drug: Neratinib at RP2D — Phase 1b: Determined dose
  Arms: Phase 1b: Platinum Resistant Expansion Cohort

SUMMARY:
To determine the recommended phase 2 dose (RP2D) of niraparib and neratinib in combination in patients with advanced solid tumors during Phase 1. To evaluate clinical benefit (≥4-month progression-free survival [PFS]) of niraparib and neratinib in patients with platinum-resistant ovarian cancer in Phase 1b.

DETAILED DESCRIPTION:
This study is a single-arm, open-label, phase 1/1b trial to determine the RP2D of neratinib and niraparib when given in combination to patients with advanced solid tumors. The RP2D will be identified during the phase 1 dose escalation portion of the study using a modified 3+3 design and evaluated in a phase 1b dose expansion cohort of up to 12 patients with platinum-resistant ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* Disease Characteristics
* Phase 1: Patients with advanced solid tumors, excluding primary CNS and prostate tumors, that have progressed during or after treatment with approved therapies or for which there is no standard effective therapy available or
* Phase 1b: Female patients with ovarian cancer who:
* Are platinum resistant (progressed within 6 months of finishing platinum therapy) and
* Have received at least 2 prior lines of therapy and
* Do not have a BRCA germline mutation
* Measurable or evaluable disease by RECIST 1.1
* Age ≥ 18 years
* ECOG performance status 0 or 1
* Adequate bone marrow function as defined below:

  * Absolute neutrophil count (ANC) ≥ 1,500/mm3
  * Platelets ≥ 100,000/mm3 (untransfused)
  * Hemoglobin ≥9 g/dL (untransfused)
* Adequate renal function as defined below:

  * Serum creatinine ≤ 1.5 x upper limit of normal (ULN) for the laboratory OR calculated
  * Or actual creatinine clearance ≥ 30 mL/min (see Appendix 2 for the Cockcroft-Gault formula for calculating creatinine clearance)
* Adequate hepatic function as defined below:

  * Total bilirubin ≤ 1.5 x ULN for the laboratory OR direct bilirubin ≤ 1.0 x ULN
  * Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN (≤ 3x ULN when liver metastases are present)
* Patients receiving corticosteroids may continue as long as their dose is stable for least 4 weeks prior to initiating protocol therapy
* Patients must agree not to donate blood during the study or for 90 days after the last dose of study treatment
* A woman of childbearing potential (WCBP) must have a documented negative serum pregnancy test within 7 days prior to initiating study treatment and agree to abstain from activities that could result in pregnancy from screening through 90 days after the last dose of study treatment. Non Childbearing potential is defined as follows (by other than medical reasons):

  * ≥45 years of age and has not had menses for >1 year
  * Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone (FSH) value in the postmenopausal range upon screening evaluation
  * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 180 days after the last dose of study treatment. Information must be captured appropriately within the site's source documents. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
* Participant must agree to not breastfeed during the study or for 30 days after the last dose of study treatment.
* Male participant agrees to use an adequate method of contraception starting with the first dose of study treatment through 90 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
* Participant must agree to not donate sperm during the study or for 90 days after the last dose of study treatment
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Any investigational agent within 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior to initiating study treatment
* Simultaneous enrollment in any other interventional clinical trial
* Active, uncontrolled diarrhea leading to dehydration or electrolyte disturbances not controlled with oral repletion
* Serious (ie, grade ≥ 3) uncontrolled infection
* Major surgery ≤ 3 weeks prior to initiating study treatment and patient must have recovered from any surgical effects.
* Radiation encompassing >20% of the bone marrow within 2 weeks, or any radiation therapy within 1 week, prior to initiating study treatment.
* Transfusion of platelets or red blood cells ≤ 4 weeks prior to initiating study treatment
* Receipt of colony-stimulating factors (e.g., granulocyte colony-stimulating factor [GCSF], granulocyte macrophage colony- stimulating factor [GM-CSF], or recombinant erythropoietin) within 4 weeks prior to initiating study treatment
* Known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
* Known brain or leptomeningeal metastasis
* Diagnosis, detection, or treatment of another type of invasive cancer ≤ 2 years prior to initiating study treatment
* Active or clinically significant cardiac disease including any of the following;

  * Unstable angina (eg, angina symptoms at rest) or onset of angina within 3 months prior to initiating study treatment
  * Myocardial infarction diagnoses within 6 months prior to initiating study treatment
  * New York Heart Association (NYHA) class III or IV congestive heart failure
  * Uncontrolled hypertension
* Inability to swallow medication
* Known hypersensitivity to niraparib or neratinib components or excipients
* Known or suspected malabsorption condition or obstruction Note: Use of pancreatic enzyme supplements is allowed to control malabsorption
* Inability to shift medications as follows:

  * Antacids (eg, calcium carbonate): dose at least 3 hours after dosing with neratinib
  * H2 receptor antagonists: dose must be taken at least 2 hours after or 10 hours before dosing with neratinib
* Planned ongoing treatment with other drugs thought to potentially have adverse interactions with either of the medications included in the study treatment:

  * Proton pump inhibitors (PPIs). Must discontinue use 10 days prior to initiating study therapy.
  * High-risk P-glycoprotein (P-gp) substrates (eg, digoxin, dabigatran).
  * Strong or moderate CYP3A4 inhibitors and/or Strong or moderate CYP3A4 inducers. Examples of clinical inhibitors and clinical inducers for P450-mediated metabolism and classification of strong, moderate, and weak interactions are available through the FDA website: http://www.fda.gov/Drugs/DevelopmentApprovalProcess/DevelopmentResources/DrugInteractionsLabeling/ucm093664.htm
  * If such medications have been used, patients must have discontinued these agents ≥ 2 weeks prior to initiating study treatment.
* Pregnancy or breastfeeding
* Medical, psychological, or social condition that, in the opinion of the investigator, may increase the patient's risk or limit the patient's adherence with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-08-24 (Actual); Primary Completion 2026-08-27 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: To determine the Recommended phase 2 dose (RP2D) of niraparib and neratinib in patients with advanced solid tumors | 4 Months
  The RP2D will be identified during the phase 1 dose escalation portion of the study using a modified 3+3 design and evaluated in a phase 1b dose expansion cohort of up to 12 patients with platinum-resistant ovarian cancer.
Phase 1b: To evaluate clinical benefit (≥4-month progression-free survival [PFS]) of niraparib and neratinib in patients with platinum-resistant ovarian cancer. | 4 months
  Phase 1b: To evaluate clinical benefit (≥4-month progression-free survival [PFS]) of niraparib and neratinib given at the RP2D to in patients with platinum-resistant ovarian cancer. To evaluate the clinical benefit, (defined as ≥4-month progression free survival (PFS), using Response Evaluation Criteria in Solid Tumors (RECIST 1.1) criteria in patients with platinum-resistant ovarian cancer.

SECONDARY OUTCOMES:
To assess the frequency of adverse events (AEs) | 5 months
  To assess adverse events (AEs) characterized and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI CTCAE V 5.0) to determine safety and toxicity of the combination of neratinib and niraparib
Preliminary efficacy (objective response rate [ORR]) of niraparib and neratinib in patients with advanced solid tumors. | 5 years
  To evaluate the objective response rate (ORR): The percentage of patients with objective response either partial response (PR) or complete response(CR), by analysis using RECIST 1.1 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Poklepovic, MD, Principal Investigator — Massey Cancer Center
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No